CLINICAL TRIAL: NCT04559165
Title: Efficacy and Safety of Sericin and Chitosan Cream for Preventing and Limiting the Progressive of Pressure Sore
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Collaborators: Police General Hospital (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Dh09066063
Record Dates: First submitted 2020-09-15; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Pressure Ulcer
MeSH Terms: conditions — Pressure Ulcer | interventions — Sericins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sericin and chitosan cream (Experimental): Apply sericin and chitosan cream on pressure ulcer 2 times/day for 21 days.
  Interventions: Other: sericin and chitosan cream
- Cavilon cream (Active Comparator): Apply cavilon cream on pressure ulcer 2 times/day for 21 days.
  Interventions: Other: sericin and chitosan cream

INTERVENTIONS:
Other: sericin and chitosan cream — sericin and chitosan cream

SUMMARY:
To evaluate efficacy and safety of sericin and chitosan cream for preventing and limiting the progressive of pressure sore in 20 patients

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years old
* 2-digit Stirling Pressure Sore Severity Scale less than or equal to 2.4
* No chitosan, sericin, and dimethicone allergy
* Without skin diseases
* Without Autoimmune diseases
* Willingness to participate

Exclusion Criteria:

* Have uncontrolled diseases
* Have complication or adverse effects during the time of participation
* Cannot follow protocol
* Pregnancy or lactation
* Participate in other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09-15 (Estimated); Primary Completion 2021-05-16 (Estimated); Study Completion 2021-06-16 (Estimated)

PRIMARY OUTCOMES:
Pressure ulcer scale for healing | 21 days
  Score 0 to 17, higher scores mean a worse outcome

SECONDARY OUTCOMES:
Erythema index | 21 days
  Erythema index will be measured using Cutometer (Mexameter). There is no unit. Higher value mean higher risk of post inflammatory reaction.
Melanin index | 21 days
  Melanin index will be measured using Cutometer (Mexameter). There is no unit. Higher value mean higher risk of post inflammatory reaction.
Transepidermal water loss | 21 days
  Transepidermal water loss index of skin will be measured using Cutometer (Tewameter). There is no unit. Higher value mean higher risk of unhealthy skin.
Moisture index | 21 days
  Moisture index of skin will be measured using Cutometer (Corneometer). There is no unit. Higher value mean lower risk of unhealthy skin.
Adverse events | 21 days
  Adverse events will be observed. They will be recorded as "present" or "not present"

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pharmacy Practice, Faculty of Pharmaceutical Sciences, Chulalongkorn Unviersity, Bangkok, Thailand